CLINICAL TRIAL: NCT00702000
Title: Clinical Determinants of Handgrip Strength in Critically Ill Adults: Pilot Study
Brief Title: Study of Intensive Care Unit (ICU)-Acquired Weakness (Handgrip Strength Study)
Status: Completed | Type: Observational
Sponsor: Naeem Ali, MD (Other)
Responsible Party: Sponsor-Investigator, Naeem Ali, MD, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2008H0081
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Peripheral Muscle Strength
Keywords: ICU acquired paresis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1.: Those with ICU-acquired weakness

SUMMARY:
To better understand ICU-acquired weakness in patients requiring mechanical ventilation in the Intensive Care Unit.

DETAILED DESCRIPTION:
We have generated the hypothesis that handgrip strength can be used to develop our understanding of the effects of critical illness on peripheral muscle strength.

To begin to develop this hypothesis, a better understanding of the determinants of handgrip strength needs to be developed. As a result we propose to perform a prospective observational study examining the clinical factors that are associated with handgrip strength. Several clinical factors are known to be associated with increased risk of developing ICUAP while hospitalized: multiple organ failure, severe sepsis, female gender and treatments like steroids. As many of these risk factors are not modifiable, the opportunity to intervene is unclear. However, by attempting to better describe the spectrum of strength deficits experienced by critically ill patients we may better be able to dissect and prevent ICUAP.

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients admitted to the Medical ICU

  * Age ≥ 18 years of age at ICU admit.
  * Requiring mechanical ventilation for at least 24 hours

Exclusion Criteria:

* • Moribund or in the process of withdrawal of life support

  * Patient, family or physicians not in favor of continued support until awakening.
  * Profound neurologic injury associated with little or no chance of awakening.
  * Active consideration of a diagnosis of brain death by treating physicians.
  * Known history of chronic neurological disease resulting in muscle weakness in more than two limbs.
  * Inability to perform handgrip dynamometry prior to acute illness.
  * Subject is a Non-english speaker
  * Subject or surrogate unable to provide informed consent.
  * ICU stay of greater than 24 hours within the last thirty days or at any point during the current hospitalization
  * Greater than seven days of hospital care prior to hospital admission.
  * Greater than five days since inclusion criteria met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects requiring prolonged mechanical ventilation in the ICU
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of performing serial assessments of strength (handgrip and limb muscle strength) in a broad population of critically ill patients. | duration of ICU stay-up to 10 days

SECONDARY OUTCOMES:
To determine the acute medical illnesses associated with weakness | duration of ICU stay-up to 10 days
To determine the modifiable risk factors associated with weakness | duration of ICU stay-up to 10 days
To determine if there is an association between handgrip strength and ICUAP risk | duration of ICU stay-up to 10 days
To generate a set of normative data for handgrip strength in critically ill patients adjusting for important non-modifiable risk factors | duration of ICU stay-up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Naeem A. Ali, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States